CLINICAL TRIAL: NCT01516697
Title: Using Thoracic Electrical Bioimpedance to Measure Stroke Volume and Cardiac Output in Patients Under Spinal Anesthesia for Cesarean Section
Brief Title: Non-invasive Cardiac Output Monitoring in Obstetric Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to enrollment subjects due to early departure of study personele
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, Assistant professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2011-P-001449
Record Dates: First submitted 2012-01-12; First posted 2012-01-25 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Complications; Cesarean Section; Anesthesia; Adverse Effect, Spinal and Epidural
Keywords: thoracic electric bioimpedance; cardiac output monitoring; cesarean section; spinal anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): The patients in Group A will serve as controls and will receive standard monitoring in addition to continuous measurement of SV and CO. The physicians will not know the CO and SV and will manage the patients in a standard fashion.
  Interventions: Procedure: Control
- experimental (Experimental): The patients in Group B will receive the same monitoring as those in Group A. But the physicians will know instantaneously the CO and SV in real time and will manage the patients accordingly.
  Interventions: Procedure: experimental

INTERVENTIONS:
Procedure: experimental — Non-invasive cardiac output monitoring using thoracic electric bioimpedance analysis via ICON® in addition of the standard monitoring during cesarean section.
  Arms: experimental
Procedure: Control — Data obtained from the non-invasive cardiac output monitor,ICON®, are not available for the anesthesia care providers.
  Arms: Control

SUMMARY:
The investigators hypothesize that continuously measuring stroke volume (SV) and cardiac output (CO) will 1) reveal hemodynamic instability in a timely manner and alert the physician promptly, 2) provide information for the physician to make the differential diagnosis as to whether the hemodynamic instability was due to vasodilatation or reduction of venous blood return, and 3) lead to appropriate and prompt treatment to improve patient outcome.

-determine the SV and CO and their kinetic change using ICON® to establish a hemodynamic profile of the patient under spinal anesthesia for cesarean section. To determine if using instantaneous measurements of SV and CO to guide patient management improves hemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45;
* receiving spinal anesthesia or combined spinal and epidural anesthesia to undergo cesarean section

Exclusion Criteria:

* Patients who have major cardiovascular disease,preexisting of hypertension or gestational hypertension, preeclampsia and body mass index greater than 35kg/m2;
* Patients who have skin lesion at the place where the electrode is supposed to be applied;
* Emergency cesarean section patients.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Maximum percentage changes in mean blood pressure after spinal anesthesia | baseline before spinal anesthesia and up to 20 minutes after spinal anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States